CLINICAL TRIAL: NCT06922240
Title: Effect of Discontinuation of Riociguat on Right Heart Function in Patients With CTEPH After Combination Therapy
Brief Title: Riociguat-Discontinue Effects on Right HEART in CTEPH (RED-HEART)
Acronym: RED-HEART
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suqiao Yang (Other)
Collaborators: China-Japan Friendship Hospital (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor-Investigator, Suqiao Yang, professor, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRWEP2024W112030108
Record Dates: First submitted 2025-03-23; First posted 2025-04-10 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic Thromboembolic Pulmonary Hypertension; Riociguat; Right heart function
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- riociguat group (Active Comparator): The subject was given comprehensive treatment in accordance with the guidelines and oral riociguat.
  Interventions: Drug: Riociguat
- routine treatment group (Experimental): The subject was given comprehensive treatment in accordance with the guidelines.
  Interventions: Drug: Routine Treatment

INTERVENTIONS:
Drug: Riociguat — On the basis of the comprehensive treatment in line with the guidelines, including conventional diuresis, anticoagulation, oxygen inhalation, etc., continue oral administration of riociguat for treatment.
  Arms: riociguat group
Drug: Routine Treatment — On the basis of the comprehensive treatment in line with the guidelines, including conventional diuresis, anticoagulation, oxygen inhalation, etc, and stop taking riociguat
  Arms: routine treatment group

SUMMARY:
Riociguat and balloon pulmonary angioplasty (BPA) are established standard-of-care interventions for inoperable chronic thromboembolic pulmonary hypertension (CTEPH) with comparable evidence levels. However, the optimal combined treatment strategy remains unclear. Specifically, there is no consensus on whether riociguat should be continued long-term after achieving hemodynamic stability with BPA. Additionally, the long-term effects of riociguat discontinuation on right ventricular (RV) structure and function remain poorly characterized, particularly due to the lack of comprehensive noninvasive evaluations integrating cardiac magnetic resonance (CMR) and echocardiography. This prospective study aims to determine the hemodynamic impact of riociguat discontinuation in inoperable CTEPH patients who have achieved BPA treatment endpoints using right heart catheterization (RHC). Evaluate RV remodeling and functional changes after riociguat cessation through multimodal noninvasive imaging (CMR, echocardiography). Assess safety outcomes and identify potential rebound pulmonary hypertension or decompensated RV dysfunction associated with riociguat withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* CTEPH was diagnosed and one of the following three factors was met: Pulmonary endarterectomy was technically impossible; Pulmonary endarterectomy is technically feasible, but the risk-benefit ratio is poor; Residual/recurrent pulmonary hypertension after pulmonary endarterectomy
* Subjects had been treated with BPA and had received a stable dose of riociguat for ≥12 weeks
* mPAP < 30mmHg
* Male subjects and female subjects of reproductive age are required to use effective contraception for at least 28 days after signing the informed consent form. Male subjects are not allowed to donate sperm and female subjects are not allowed to breastfeed.
* Subjects voluntarily sign written informed consent

Exclusion Criteria:

* Severe hepatic and renal insufficiency (Child-Pugh Grade C/creatinine clearance < 30ml/min·1.73m²)
* The presence of severe infectious disease or severe bleeding tendency
* Combined with pulmonary hypertension of other types than CTEPH
* Other pulmonary hypertension targeting drugs are being used
* The expected survival time with cancer or other diseases is less than 6 months
* Pregnancy, lactation
* Subjects are currently participating in an interventional clinical trial
* In the investigator's judgment, a subject's medical abnormality, physical condition, or medical history may affect his or her ability to participate in or complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Cardiac Output at 6 Months. | Baseline and 6-month follow-up
  Cardiac Output was measured by right heart catheterization.

SECONDARY OUTCOMES:
Change from Baseline in the Pulmonary Vascular Resistance at 6 Months. | Baseline and 6-month follow-up
  Pulmonary Vascular Resistance was measured by right heart catheterization.
Change from Baseline in the concentration of NT-proBNP at 6 Months. | Baseline and 6-month follow-up
  The concentration of NTproBNP in serum was detected in pg/ml
Change from Baseline in the 6-minute walking distance at 6 Months. | Baseline, 3-month follow-up, and 6-month follow-up
  6-minute walking distance was measured by 6-minute walking test
All-cause mortality | From the baseline to the completion follow-up,an average of 6 months
  Observe and record All-cause mortality
Combined incidence of all-cause death, re-hospitalization or disability/incapacity events due to clinical exacerbation of pulmonary hypertension | From the baseline to the completion follow-up,an average of 6 months
  Observe and record All-cause mortality, clinical exacerbation of pulmonary hypertension leading to re-hospitalization or disability/incapacity

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Chao-Yang Hospital, Beijing, China
  - China-Japan Friendship Hospital, Beijing, China
  - Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No